# **TUNG WAH COLLEGE**

#### **Informed Consent Form for Adult**

# **Evaluation of Balance and Gait Weight Distribution in Patients with Vertebral Column Fractures**

You are invited to participate in a research study conducted by Dr. Anthony Kwok in the School of Medical and Health Sciences at Tung Wah College (TWC).

## PURPOSE OF THE STUDY

The purpose of the study is to identify the association of balance and gait weight distribution with fall risk in patients with vertebral column fractures.

## **PROCEDURES**

Participants will be interviewed with a set of questionnaires regarding your functionality in activities in daily living, and assessed for the balance performance and gait weight distribution under the supervision of research assistants. This will involve a 2-hours visit to the College for the interview and assessments. The procedure will not be video-recorded / audio-recorded.

## POTENTIAL RISKS / DISCOMFORTS AND THEIR MINIMIZATION

The assessments are of low impact and low risk. These will be performed under the supervision of a registered physiotherapist and research assistants to minimize the potential risks and discomforts.

Participants can seek help from the registered physiotherapist and research assistants in case of any bad effects of the procedure.

## **COMPENSATION FOR PARTICIPATION**

The participation is on voluntarily basis. No compensation is given for the participation.

# POTENTIAL BENEFITS

This research does not provide you with personal benefits, but the data collected will provide valuable information for studying the vertebral column fractures.

# **CONFIDENTIALITY**

All information obtained will be used for research purposes only. Subject will not be identified by name in any report of the completed study.

# DATA RETENTION

All the information collected for this research will be kept confidential. Information collected for this research will only be accessible by the principal investigator and the research assistants, and will be discarded properly within 5 years after the research report is presented.

# PARTICIPATION AND WITHDRAWAL

This study follows the Declaration Helsinki. Your participation is voluntary. This means that you can choose to stop at any time without negative consequences.

# **QUESTIONS AND CONCERNS**

If you have any questions or concerns about the research, please feel free to contact Dr. Anthony Kwok at 852-3468 6670. If you have questions about your rights as a research subject, contact the Secretary, Research Ethics Committee (REC), TWC (ro@twc.edu.hk).

| SIGNATURE | |
|---|---|
| I | (Name of Subject) |
| understand the procedures described above and agree to par | rticipate in this study. |
| I ** wish / do not wish to be identified. | |
| (** Please delete as appropriate.) | |
| | Signature: |
| | Date: |